CLINICAL TRIAL: NCT04262674
Title: Development of an Innovative, Non-invasive, Wearable Multi-parameter System for the Early Prediction of Cognitive Decline and Dementia in Older Adults
Brief Title: Non-invasive, Wearable Multi-parameter System for the Early Prediction of Cognitive Decline and Dementia in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Empa, Swiss Federal Laboratories for Materials Science and Technology (Other)
Collaborators: Geriatrische Klinik St. Gallen (Other); ETH Zurich (Other)
Responsible Party: Principal Investigator, Patrick Eggenberger, Principal Investigator, Postdoc, Empa, Swiss Federal Laboratories for Materials Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 5213.00187
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Mild Cognitive Impairment; Healthy Aging
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-motor training (Experimental): Simultaneous cognitive-motor training (i.e. exergame) and strength training
  Interventions: Other: Cognitive-motor training
- Control (No Intervention): Passive control group

INTERVENTIONS:
Other: Cognitive-motor training — Simultaneous cognitive-motor training and strength training
  Other Names: Exergame; Step Mania
  Arms: Cognitive-motor training

SUMMARY:
This project develops an innovative screening system and prediction model to detect preclinical symptoms of cognitive impairment and predict the potential development of mild cognitive impairments and dementia in older adults. The earliest possible detection of preclinical symptoms is prerequisite to improve the efficacy of subsequent preventative non-pharmacological, life-style and exercise related, personalized treatment interventions.

DETAILED DESCRIPTION:
BACKGROUND: Early detection of preclinical symptoms and prediction of potential development of mild cognitive impairment (MCI) and Alzheimer's disease (AD) could improve non-pharmacologic, life-style and exercise related preventative interventions' efficacy and slow-down disease progression. To achieve this goal, discriminating the earliest preclinical stage of MCI/AD from healthy state would be necessary. However, this is still challenging and current clinical methods are not feasible for preventative screening in larger populations of older adults, as they involve invasive sampling of molecular blood or cerebrospinal fluid biomarkers, as well as expensive brain imaging and extensive neuropsychological testing. Recently, several non-invasive alternative measures, including electroencephalography (EEG), gait analysis, heart rate variability (HRV), and core body temperature (Tc), were shown to be associated with preclinical symptoms of MCI/AD and to predict disease progression.

AIM: The investigators aim to combine these measures in a novel non-invasive multi-parameter prediction model, which better reflects multimodal symptomatology compared to currently used methods and, therefore, allows discriminating healthy persons from MCI state with adequate sensitivity (i.e. >80%).

METHODS: A cohort of 85 older adults, ≥65 years of age, including healthy persons and patients with MCI, will be recruited. Assessments will be performed at baseline, after 2 months (within these two 2 months one group will follow a cognitive-motor training intervention, while the other serves as passive control), and at 12-month follow-up. Assessments include EEG, gait analysis, HRV, and Tc at rest and during walking, and will be compared to reference measures of MCI status, including neuropsychological tests, to develop the prediction model and evaluate its sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* participants have to be older than 65 years of age
* cognitively healthy or diagnosed with MCI
* able to walk at least 8 minutes for gait analysis, with or without walking aids
* live independently or in a retirement home (classified 0, 1, or 2 within the Swiss classification system for health-care requirements BESA-levels [German abbreviation for: Bewohner-Einstufungs- und Abrechnungs-System; level 0 meaning the person does not need care or treatment; level 1 to 2 meaning, the person only needs little care or treatment])
* sign informed consent

Exclusion Criteria:

* previously diagnosed dementia, e.g. Alzheimer's disease
* recent head injury
* judgment by the participant's primary care physician will be required in the case of acute or instable chronic diseases (e.g. stroke, diabetes) and rapidly progressing or terminal illnesses

Additional exclusion criteria for the subgroup of 15 participants who would agree to take the telemetric gastrointestinal temperature pill:

* history of operations and/or disease related to the gastrointestinal tract within last 5 years
* implanted medical device
* planned MRI examination
* nausea, vomiting, constipation or abdominal pain within 1 months prior to the day of planned measurement

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Electroencephalography (EEG) | 30 minutes
  EEG frequency bands (Hz) will be assessed during 10 minutes at rest in a seated position (5 min eyes closed, 5 min eyes open) and will be recorded using a wearable system covering the frontal, parietal, temporal, and occipital cortex and integrating 20 gel-pad electrode channels. The assessment will be continued during the subsequent gait protocol which consists of 8 minutes of walking back and forth at preferred speed on a 20 m track.
Gait speed analysis with inertial sensors | 15 minutes
  The gait protocol consists of 8 minutes of walking back and forth at preferred speed on a 20 m track. Thereby, walking speed (m/s) will be assessed using inertial sensors attached to the feet.
Gait variability analysis with inertial sensors | 15 minutes
  The gait protocol consists of 8 minutes of walking back and forth at preferred speed on a 20 m track. Thereby, step length variability (%) and step time variability (%) will be assessed using inertial sensors attached to the feet.
Heart rate variability (HRV) indices SDNN and RMSSD with two-lead electrocardiogram chest belt | 10 minutes
  The HRV indices SDNN (ms) and RMSSD (ms) will be assessed during 10 minutes in a seated position, using a two-lead electrocardiogram chest belt.
Heart rate variability (HRV) index HF power with two-lead electrocardiogram chest belt | 10 minutes
  The HRV index HF power (ms^2) will be assessed during 10 minutes in a seated position, using a two-lead electrocardiogram chest belt.
Body temperature (T) with temperature sensors (thermistors) | 30 minutes
  T will be assessed under controlled climatic conditions (22°C/40% relative humidity) measuring skin T (°C) at the scapula and the the ribs (lateral) using temperature sensors (thermistors) during 10 minutes sitting and 8 minutes walking as described above.

SECONDARY OUTCOMES:
Cognitive performance with neuropsychological tests | 1 hour
  Neuropsychological tests will be performed to assess general cognitive performance (Quick Mild Cognitive Impairment screen), episodic memory (associative memory, Face-Name Associative Memory Exam, FNAME-12 test), semantic verbal fluency (category and letter fluency test), and executive functions (Trail Making Tests A/B, Stroop Test). The score of each test will be standardized and added up into a combined score of cognitive performance (z-score).
Core body temperature (Tc) with telemetric gastrointestinal temperature pill | 16 hours
  In a subgroup of 15 participants, Tc (°C) will be recorded with a telemetric gastrointestinal temperature pill over a period of 16 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Eggenberger, Dr., Principal Investigator — Empa, Swiss Federal Laboratories for Materials Science and Technology
Locations (1):
- Empa, Sankt Gallen, Canton of St. Gallen, Switzerland